CLINICAL TRIAL: NCT03755388
Title: Long-term Prospective Interventional Clinical Trial of an MRI Based Patient Specific Focal Knee Resurfacing Implant
Brief Title: Clinical Trial of an MRI Based Patient Specific Focal Knee Resurfacing Implant
Acronym: Episealer2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S61896
Record Dates: First submitted 2018-11-05; First posted 2018-11-28 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Cartilage Damage; Knee Injuries
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Episealer group (Experimental): Subjects with a focal cartilage lesion of the distal femur in which biological surgical methods have failed or are not eligible
  Interventions: Device: Episealer

INTERVENTIONS:
Device: Episealer — Placing Episealer device

SUMMARY:
The goal of this study is to evaluate the efficacy, safety and performance of the Episealer® device in a sample size of 30 patients and on the long term (10 years follow-up).

DETAILED DESCRIPTION:
Lesions in the cartilage are common disorders. In the knee, cartilage lesions are found in over 50 % of all arthroscopies, where 25 % of these are of focal character and the majority are found in the medial femoral condyle. The quality of life of patients with focal cartilage defects is significantly affected and it has been shown that the quality of life is affected to the same extend as in patients scheduled for knee replacement. Arthroscopy lavage and debridement micro fracturing, mosaic plasticity as well as osteochondral autograft transplantation (OATS) are methods used for treatment of the lesions. Some have shown to help the patients but there is an ongoing treatment gap especially for patients with knee lesions and early osteoarthritis.

Episurf Medical has developed a Focal Knee Resurfacing (FKR) implant, the Episealer® implant. The implant is used for treatment of focal cartilage lesions of the lateral or medial femoral condyle in order to alleviate pain and improve range of motion. The implant and surgical instruments are customized to each patient's joint anatomy, position, and size of injury, based on patient-specific images (MRI). The Episealer® device is CE marked.

The Episealer® implant consists of a peg and a hat. The implant exists in five different diameters (12,14,17, 20 and 25mm), depending on the lesion size. The shape of the hat is circular or oval.

The Episealer® implant is made of biocompatible cobalt/chromium/molybdenum alloy. To enhance the osseointegration, the implant is coated with biocompatible hydroxyapatite onto an interlaying biocompatible pure titanium coating.

A previous study (S57685) showed that Episealer is a viable option for focal cartilage lesions of the distal femur not responding, or not eligible for, biological treatment options (eg. microfracturing). This device is a good solution when there are no alternative treatments, except prosthesis surgery, available.

The goal is to evaluate the efficacy, safety and performance of the Episealer® device in a larger sample size and on the long term.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a focal cartilage lesion of the distal femur in which biological surgical methods have failed or are not eligible
* Minimal age 18 years (Preferred age group >40 years)
* Suitable for implant, to be determined by analysis of MRI imaging. Suitability is set by the size and location of the lesion.
* Informed consent

Exclusion Criteria:

* Under age (<18yrs)
* Active or recent (<1 yr) septic arthritis of the involved knee
* Associated symptomatic untreated ligamentary or meniscal pathology in the involved knee
* (Severe) osteoarthritis in the involved or other compartments of the involved knee
* Severe osteoporosis
* MRI not possible (eg. due to pacemaker)
* Marked valgus- or varus alignment (>6 degrees)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-09-20 (Actual); Primary Completion 2034-12 (Estimated); Study Completion 2034-12 (Estimated)

PRIMARY OUTCOMES:
Survival | 10 years
  Presence of the implant in the patient up to 10 years post treatment with loss/revision of the primary implant as endpoint

SECONDARY OUTCOMES:
Radiographic measurements | 10 years
  Efficacy will be evaluated with the comparison of the pre- and post- operative radiographs
Knee injury and Osteoarthritis Outcome Score (KOOS) | 10 years
  Performance will be evaluated with the comparison of the pre- and post- operative KOOS-scores. Scoring: each item is scored between 0 and 4 and the raw score of each section is the sum or item scores. The score is then converted into a 0-100 scale. A higher score indicates fewer problems
Visual Analogue Scale (VAS) pain | 10 years
  Performance will be evaluated with the comparison of the pre- and post- operative VAS-scores. Score between 0 and 10. Higher score indicates more pain.
Complications | 10 years
  Safety will be evaluated by monitoring AEs, unanticipated device effects and subsequent interventions through 10 years post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Hilde Vandenneucker, MD, PhD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No